CLINICAL TRIAL: NCT03088306
Title: Comparative Effectiveness of Multi-modal Pain Management Versus Standard Intra- and Post-operative Analgesia: Randomized Controlled Clinical Trial to Reduce Post-operative Pain and Opioid Use Among Patients Undergoing Lumbar Spine Surgery
Brief Title: Improving Pain and Reducing Opioid Use (IPaRO) in Lumbar Spine Surgery Patients
Acronym: IPaRO
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: North American Spine Society (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00113816
Record Dates: First submitted 2017-02-22; First posted 2017-03-23 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Lumbar Spinal Stenosis; Lumbar Spinal Instability; Lumbar Spine Degeneration
MeSH Terms: conditions — Spinal Stenosis | interventions — Oxygen; Hydromorphone; Fentanyl; Acetaminophen; Gabapentin; Diazepam

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard analgesia use (Active Comparator): A strategy to manage pain in the peri-operative period that is in common clinical use.
  Interventions: Drug: Standard analgesia use [Oxygen]; Drug: Standard analgesia use [Hydromorphone]; Drug: Standard analgesia use [Volatile Anesthesia]; Drug: Standard analgesia use [Fentanyl]
- Multi-modal pain management (Active Comparator): A strategy to manage pain in the peri-operative period that is in common clinical use that is designed to reduce the need for post-operative opioid medication.
  Interventions: Drug: Multi-modal pain management [Acetaminophen + Gabapentin]; Drug: Multi-modal pain management [Fentanyl]; Drug: Multi-modal pain management [Intravenous Ketamine]; Drug: Multi-modal pain management [Valium + Gabapentin]

INTERVENTIONS:
Drug: Standard analgesia use [Oxygen] — A protocol directed and clinically appropriate post-operative analgesia. In this study, standard post-operative analgesia is defined as: oxygen, volatile anesthesia, fentanyl, hydromorphone.
  Arms: Standard analgesia use
Drug: Standard analgesia use [Hydromorphone] — A protocol directed and clinically appropriate post-operative analgesia. In this study, standard post-operative analgesia is defined as: oxygen, volatile anesthesia, fentanyl, hydromorphone.
  Arms: Standard analgesia use
Drug: Standard analgesia use [Volatile Anesthesia] — A protocol directed and clinically appropriate post-operative analgesia. In this study, standard post-operative analgesia is defined as: oxygen, volatile anesthesia, fentanyl, hydromorphone.
  Arms: Standard analgesia use
Drug: Standard analgesia use [Fentanyl] — A protocol directed and clinically appropriate post-operative analgesia. In this study, standard post-operative analgesia is defined as: oxygen, volatile anesthesia, fentanyl, hydromorphone.
  Arms: Standard analgesia use
Drug: Multi-modal pain management [Acetaminophen + Gabapentin] — Administration of acetaminophen (1 gm po) plus gabapentin (600-1200 mg po) in the preparation area prior to surgery; pre-induction opioid titration with fentanyl until pain is relieved and/or respiratory depression ensues; intravenous ketamine (1 mg/kg load prior to incision then 10 mcg/kg/min) during surgery; acetaminophen, valium plus gabapentin during hospitalization; and prescription for acetaminophen, valium plus gabapentin at discharge.
  Arms: Multi-modal pain management
Drug: Multi-modal pain management [Fentanyl] — Administration of acetaminophen (1 gm po) plus gabapentin (600-1200 mg po) in the preparation area prior to surgery; pre-induction opioid titration with fentanyl until pain is relieved and/or respiratory depression ensues; intravenous ketamine (1 mg/kg load prior to incision then 10 mcg/kg/min) during surgery; acetaminophen, valium plus gabapentin during hospitalization; and prescription for acetaminophen, valium plus gabapentin at discharge.
  Arms: Multi-modal pain management
Drug: Multi-modal pain management [Intravenous Ketamine] — Administration of acetaminophen (1 gm po) plus gabapentin (600-1200 mg po) in the preparation area prior to surgery; pre-induction opioid titration with fentanyl until pain is relieved and/or respiratory depression ensues; intravenous ketamine (1 mg/kg load prior to incision then 10 mcg/kg/min) during surgery; acetaminophen, valium plus gabapentin during hospitalization; and prescription for acetaminophen, valium plus gabapentin at discharge.
  Arms: Multi-modal pain management
Drug: Multi-modal pain management [Valium + Gabapentin] — Administration of acetaminophen (1 gm po) plus gabapentin (600-1200 mg po) in the preparation area prior to surgery; pre-induction opioid titration with fentanyl until pain is relieved and/or respiratory depression ensues; intravenous ketamine (1 mg/kg load prior to incision then 10 mcg/kg/min) during surgery; acetaminophen, valium plus gabapentin during hospitalization; and prescription for acetaminophen, valium plus gabapentin at discharge.
  Arms: Multi-modal pain management

SUMMARY:
Patients presenting for lumbar spine surgery experience pain related to their spine condition. Following surgery, these patients also experience surgical pain resulting from disruption of skin, muscle tissue, vertebrae, intervertebral discs, and facet joints. This pain is often treated with opioid medications - with roughly 40% of patient experiencing sub-optimal pain management. Adequate pain control has become a top priority among professional societies, healthcare systems, and accrediting agencies. The current proposal will provide this critical evidence of feasibility and acceptability of a multi-modal pain management plan for patients undergoing lumbar spine surgery. Additionally, this study will provide critical preliminary data to compare the effectiveness of protocol-driven multi-modal pain management to control post-operative pain, reduce opioid medication use, and improve physical activity, sleep, and health.

DETAILED DESCRIPTION:
Patients presenting for lumbar spine surgery experience pain related to their spine condition. Following surgery, these patients also experience surgical pain resulting from disruption of skin, muscle tissue, vertebrae, intervertebral discs, and facet joints. Proper pain management is necessary to reduce pain-related and medication side effects and to promote rehabilitation. This pain is often treated with opioid medications - with roughly 40% of patient experiencing sub-optimal pain management. Adequate pain control has become a top priority among professional societies, healthcare systems, and accrediting agencies.

Multi-modal pain management strategies have been proposed to (1) control pre-operative pain related to spine pathology; (2) employ non-opioid medication peri-operatively to pre-empt post-operative surgical pain; and (3) monitor and control pain intensity before and after surgery. There is a demonstrated lack of evidence regarding optimal post-operative protocols and pathways. The investigators have planned a randomized clinical trial to compare the effectiveness of two methods of peri-operative pain management to reduce post-operative pain and opioid use among patients undergoing lumbar spine surgery.

Prior to submission to National Institutes of Health (NIH), Agency for Healthcare Research and Quality (AHRQ), or Patient Centered Outcomes Research Institute (PCORI), it is necessary to demonstrate the feasibility and acceptability of the trial protocol. The current proposal will provide this critical evidence of feasibility and acceptability of a multi-modal pain management plan for patients undergoing lumbar spine surgery. Additionally, this study will provide critical preliminary data to compare the effectiveness of protocol-driven multi-modal pain management to control post-operative pain, reduce opioid medication use, and improve physical activity, sleep, and health.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants will be English-speaking adults who are presenting to a spine surgeon (orthopaedic or neurosurgeon) for surgical treatment of a lumbar degenerative condition (spinal stenosis, spondylosis with or without myelopathy, and degenerative spondylolisthesis) using laminectomy with or without arthrodesis (i.e. fusion).

Exclusion Criteria:

* A microsurgical technique as the primary procedure, such as an isolated laminotomy or microdiscectomy.
* Spinal deformity as the primary indication for surgery.
* Spine surgery secondary to pseudarthrosis, trauma, infection, or tumor.
* Back and/or lower extremity pain < 3 months indicating no history of sub-acute or chronic pain.
* History of neurological disorder or disease, resulting in moderate to severe movement dysfunction.
* Presence of schizophrenia or other psychotic disorder.
* Patient refusal to participate.
* Known allergic reactions to any of the study medications
* Surgery under a workman's compensation claim.
* Not able to return to clinic for standard follow-up visits with surgeon.
* Unable to provide a stable address and access to a telephone.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Number of participants undergoing lumbar spine surgery with complete follow-up | 52 week
  Number of participants undergoing lumbar spine surgery with complete follow-up

SECONDARY OUTCOMES:
Patient controlled analgesia (PCA) pump use | during surgical hospitalization, up to 12 weeks
  Total morphine equivalent of opioids administered by the PCA pump
Opioid medication use | up to 90 days
  How many patients were prescribed and using opioid medication over the 90 days after hospital discharge?
Patient Reported Outcomes Measurement Information System (PROMIS) Pain | at 6 and 12 weeks
  Measure of pain intensity; Range 0 - 100; Population mean 50, standard deviation 10
PROMIS Physical Function | at 6 and 12 weeks
  Measure of physical function; Range 0 - 100; Population mean 50, standard deviation 10
PROMIS Fatigue | at 6 and 12 weeks
  Measure of fatigue; Range 0 - 100; Population mean 50, standard deviation 10
PROMIS Anxiety | at 6 and 12 weeks
  Measure of anxiety; Range 0 - 100; Population mean 50, standard deviation 10
PROMIS Depression | at 6 and 12 weeks
  Measure of depression; Range 0 - 100; Population mean 50, standard deviation 10
PROMIS Sleep Disturbance | at 6 and 12 weeks
  Measure of sleep disturbance; Range 0 - 100; Population mean 50, standard deviation 10
PROMIS Satisfaction with Social Roles | at 6 and 12 weeks
  Measure of satisfaction with social roles; Range 0 - 100; Population mean 50, standard deviation 10
Health status (Medical Outcome Study Short Form 12, version 2) | at 6 and 12 weeks
  Measure of physical and mental health; Range 0 - 100; Population mean 50, standard deviation 10
Oswestry Disability Index (ODI) | at 6 and 12 weeks
  Measure of pain-related disability; Range 0% - 100%; Scores greater than 30% indicative of moderate pain-related disability

CONTACTS AND LOCATIONS:
Overall Officials: Richard L Skolasky, ScD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No